CLINICAL TRIAL: NCT03088579
Title: Intraoperative Brachytherapy for Central Nervous System Lesions: A Validation Study of a Radioactive Seed Loading Device
Status: Completed | Type: Observational
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Arizona Commerce Commission, Phoenix AZ (Unknown); GT Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 13RT022
Record Dates: First submitted 2017-03-01; First posted 2017-03-23 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Central Nervous System Lesion
Keywords: radiation shielding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: GammaTile seed loader — Patients are chosen based on symptomatic tumor/radiographic finding of a surgically accessible mass. Surgery will be done in usual fashion. A cavity will be left where the tumor was. Size of operative bed will be measured using a surgical dissector and standard operating room ruler. A sheet of surgical fabric may be used to estimate size of cavity. If pathology is positive the study treatment will continue. If not, patient will not be on trial. If patient is eligible, radiation oncologist will form custom implants using a seed(s) of Cesium-131, with other biocompatible materials used to achieve maximum dosimetric conformality. Surgeon will place constructs into cavity until the operative bed is fully addressed. Implant is not expected to migrate. Surgicel, bioglue or similar material may be used to secure seeds. Wound will be closed in standard fashion. The last 10 patients will be asked to participate in an effort to gauge costs related to radiation portion of treatment.

SUMMARY:
The researchers recognized the possible clinical usefulness of a shielded device or jig to help increase the accuracy but decrease the time of loading the seeds into the biocompatible material used intra-operatively. Therefore, the researchers created a prototype of a device called the GammaTile (GT) loader (design patent pending). The reusable device will be made of surgical quality stainless steel of sufficient thickness (greater than 10 half-value layers (HVL) to provide significant staff and user shielding as well as allowing it to be sterilized. It is utilized intraoperatively but off of the operative field and has no direct patient contact. Currently two sizes are planned. The first will accommodate a 2 inch x 2 inch collagen square and the second will accommodate a 1 inch x 1 inch collagen square. These are the most commonly used sizes of lyophilized collagen used in the Barrow Neurosurgical Institute (BNI) operating rooms (OR).

DETAILED DESCRIPTION:
This is a 100 patient observational-design study for the purpose of testing the seed loader device as a method of arranging and securing the seeds in a carrier in a set pattern for the convenient use of the neurosurgeon against the backdrop of a hodgepodge of currently available techniques (seed in suture, seed in mesh, loose seeds), all of which currently need to be secondarily secured with some additional, not currently standardized material, in a cumbersome, time-consuming, and not assuredly accurate manner. An additional primary objective will be an assessment of the loader device as a radiation protection tool for the user and staff during seed placement in the carrier and prior to intracranial carrier placement. Secondary objectives will be conformality of pre- and post-implant dosimetry (expected vs achieved) and post implant stability (seed shift) over time as judged on a routine follow up MRI. An additional proposed endpoint is an economic (cost) comparison to other modalities.

Eligible patients are those deemed appropriate for and scheduled to undergo adjuvant brachytherapy of the central nervous system as determined by the radiation oncologist and neurosurgeon. Potential candidates will have a lesion(s) that may be newly diagnosed or recurrent, in need of gross total or near gross total resection, and such that in the opinion of the operating surgeon it would be both amenable to and in need of the proposed treatment. Informed consent will be obtained. Radiation oncologist and neurosurgeon will determine appropriateness of the proposed procedure and the radiation oncologist and neurosurgeon will determine the volume and configuration of the area to be implanted.

A carrier using currently available material (lyophilized bovine-derived collagen, Duraform or similar) stocked in the BNI OR. The isotope (seeds) are also already approved for use anywhere in the body, are in use and on the hospital's radioactive materials license (RML). Patients will have pre- and post-operative computerized tomography (CT) or magnetic resonance imaging (MRI) as routine care, and post-operative CT's as per routine implant case dosimetry. All applicable radiation safety procedures will continue to be followed. The sterilizable loader(s) will be provided as a non-charge-item, and are anticipated to be classified as a "Class 1" device by the FDA as they are not implanted and have no direct patient contact.

ELIGIBILITY:
Inclusion Criteria:

* Planned for resection of aggressive primary or metastatic brain tumor and appropriate for adjuvant radiotherapy.
* Zubrod Performance Score of 0-2.
* 18 years of age or older.
* Pre-operative stereotactic CT or MRI.
* Life expectancy >26 weeks.
* History and physical for all patients and detailed neurological exams.
* Signed study-specific informed consent form prior to study entry.

Exclusion Criteria:

* Negative biopsy if presumed diagnosis on imaging.
* External beam therapy is allowed if the implant is being used instead of a boost or cone down treatment.
* Life expectancy < 26 weeks.
* Inability to undergo post-operative CT for implant assessment, or postoperative follow-up imaging.
* Major medical or psychiatric illness, which, in the investigator's opinion, would prevent completion of treatment and/or interfere with follow-up.
* Inability or refusal to provide informed consent.
* Prior radiation therapy in excess of 100Gy to site of implant.
* Patients in which there is no cranium in place (for example, bone flap removed for infection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults of either gender having a central nervous system lesion (high grade primary brain tumor and electing intra-operative brachytherapy. Participants will be patients of Barrow Brain and Spine neurosurgery group located in Phoenix AZ.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-04-02 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
User's Experience | Immediately post-operatively
  Analyze users' (radiation oncologists and neurosurgeons) experience with the loader methodology by utilizing a standardized questionnaire recording 1) time added to case, 2) the size and size range of implants utilized, 3) conformality to operative bed, and 4) ease of use. Both perceptual (subjective) and numerical (objective) data will be obtained.
Shielding | Immediately post-operatively
  Evaluate shielding (radiation protection ability) of shielded loader through mRm measurements while seeds are in loader prior to implantation: surface of loader (mRm/hour), at 1 meter (mRm/hour), and at 3 meter (mRm/hour).

SECONDARY OUTCOMES:
Post-Implant Dosimetric Analysis | Post-operative Day 1
  Using Advisory Committee on the Medical Uses of Isotopes (ACMUI) guidelines, analyze the post-implant dosimetry and compare with the pre-plan dosimetry (expected vs achieved dosimetry) both of which are standard procedures for brachytherapy.
Seed Migration | Post-operative Day 1
  Presence or absence of source (seed) migration on subsequent scans ordered for routine follow-up.
Economic Impact | Post-Operative Day 1, at follow-up per routine care (up to 5 years)
  For all study patients obtain sufficiently detailed, global costs for treatment to be able to analyze the overall cost of this modality compared to existing literature data for other forms of adjuvant therapies where available.
Progression Free Survival (PFS) | Pre-Operative and at follow-up per routine care (up to 5 year)
  The length of time during and after treatment that the participant lives with the disease but it does not get worse.
Overall Survival (OS) | Pre-Operative and at follow-up per routine care (up to 5 year)
  The length of time from when consent is signed that participants are still alive.
Zubrod Performance Scale | Pre-Operative, Post-Operative Day 1, at follow-up per routine care (up to 5 years)
  Participants ability to carry out activities of daily living will be scored per the following scale:
  0 Fully active, able to carry on all predisease activities without restriction (Karnofsky 90-100);
  1. Restricted in physically strenuous activity but ambulatory and able to carry work of a light or sedentary nature. For example, light housework, office work (Karnofsky 70-80);
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours (Karnofsky 50-60);
  3. Capable of only limited self-care, confined to bed or chair 50% or more of waking hours (Karnofsky 30-40);
  4. Completely disabled. Cannot carry on self-care. Totally confined to bed or (Karnofsky 10-20);
  5. Death (Karnofsky 0).
Neurologic Function Status Scale | Pre-Operative, Post-Operative Day 1, at follow-up per routine care (up to 5 years)
  Participants' neurologic status will be scored per the following scale:
  0 No neurologic symptoms - fully active at home/work without assistance;
  1. Minor neurologic symptoms - fully active at home/work without assistance;
  2. Moderate neurologic symptoms - fully active at home/work but requires assistance;
  3. Moderate neurologic symptoms - less than fully active at home/work and requires assistance;
  4. Severe neurologic symptoms - totally inactive requiring complete assistance at home or in institution--unable to work.

CONTACTS AND LOCATIONS:
Overall Officials: David G Brachman, MD, Study Chair — Barrow Neurological Institute; Peter Nakaji, MD, Study Chair — Barrow Neurological Institute
Locations (2):
- United States (2):
  - Barrow Brain and Spine, Phoenix, Arizona
  - Barrow Neurological Institute at St. Joseph's Hospital and Medical Center, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinnaduwage DS, Srivastava SP, Yan X, Jani S, Brachman DG, Sorensen SP. Dosimetric Impacts of Source Migration, Radioisotope Type, and Decay with Permanent Implantable Collagen Tile Brachytherapy for Brain Tumors. Technol Cancer Res Treat. 2022 Jan-Dec;21:15330338221106852. doi: 10.1177/15330338221106852. PMID 35712977